CLINICAL TRIAL: NCT04671329
Title: A Prospective, Multi-site Clinical Study to Collect User Feedback Using Affirm® Contrast Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-03
Record Dates: First submitted 2020-12-01; First posted 2020-12-17 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
Keywords: Breast Biopsy, Contrast Biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Affirm Contrast Biopsy (Other): Women 40 years of age or older recommended for biopsy who have had a suspicious finding on previous contrast enhanced imaging or have lesions that may be occult under other modalities
  Interventions: Device: Affirm Contrast Biopsy procedure

INTERVENTIONS:
Device: Affirm Contrast Biopsy procedure — Contrast Enhanced Digital Mammography (CEDM) is an extension of the existing indication for diagnostic mammography with the Selenia Dimensions system and 3Dimensions system. Biopsy targeting can be done on captured contrast enhanced images (scout and stereo pair). The CEDM application shall enable contrast enhanced breast imaging using a dual energy technique. This imaging technique can be used as an adjunct following mammography and/or ultrasound exams to localize a known or suspected lesion. Affirm Contrast Biopsy is intended for patients recommended for biopsy who have had a suspicious finding on previous contrast enhanced imaging or have lesions that may be occult under other modalities.

SUMMARY:
Currently, if a radiologist finds a suspicious lesion seen only on a diagnostic Contrast Enhanced Digital Mammography (CEDM) exam requiring biopsy the biopsy procedure would likely be performed with MRI guidance because there are currently limited solutions to biopsy with CEDM guidance. Affirm Contrast Biopsy will provide an additional solution to biopsy/localize lesions found by using a CEDM imaging modality.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 40 years of age or older recommended for biopsy who have had a suspicious finding on previous contrast enhanced imaging or have lesions that may be occult under other modalities
* Subject is able to read, understand, and sign the study specific informed consent form after the nature of the study has been fully explained to them

Exclusion Criteria:

* Subjects who require a Legally Authorized Representative (LAR) for Informed Consent
* Subjects who, based on the physician's judgement, may be at increased risk for complications associated with renal function, anticoagulant therapy, or bleeding disorders
* Subjects who have had a previous allergic reaction to IV contrast agent

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-08-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mayo Clinic, Phoenix, Arizona
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Affirm Contrast Biopsy
Started | 67
Completed | 60
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Affirm Contrast Biopsy
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Technical Success
Description: Technical success was defined as successfully completing the breast biopsy procedure with the Affirm Contrast Biopsy system for each participant (60 participants equals 60 procedures).
Time Frame: Up to 1h (time to complete the procedure)
Population: Women of 40 years of age or older that were recommended for biopsy who have had a suspicious finding on previous contrast-enhanced imaging or have lesions that may be occult under other modalities.
Measure: Count of Participants; unit: Participants
Arm/Group | Affirm Contrast Biopsy
Number analyzed (Participants) | 60
Participants | 60

ADVERSE EVENTS:
Time Frame: Up to 1h (time to complete procedure per participant)
Arm/Group | Affirm Contrast Biopsy
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

LIMITATIONS AND CAVEATS:
No limitations or caveats were found for this study. A total of 67 subjects were enrolled and seven subjects were withdrawn by the Investigator (did not complete the biopsy procedure), for a final total of 60 subjects who were included in the final analysis. The seven withdrawal cases were not related to any procedure failure but related to no lesion enhancement found or no biopsy needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/29/NCT04671329/Prot_SAP_ICF_001.pdf